CLINICAL TRIAL: NCT06540131
Title: The Impact of Ethyle Alcohol Contact Time on Corneal Epithelial Healing in Cases of Photorefractive Keratectomy
Brief Title: Studying the Effect of Ethanol Applied on the Corneal Surface During PRK Surgery.
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ismail Omar, Associate professor of ophthalmology, Minia University
Other Study IDs: 1093/03/2024
Record Dates: First submitted 2024-07-23; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Corneal Ulcer of Bilateral Eyes
Keywords: PRK; ethanol; corneal ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group of 15 seconds ethanol: Group of eyes with ethanol applied on the corneal surface for 15 seconds
- group of 30 seconds ethanol: Group of eyes with ethanol applied on the corneal surface for 30 seconds

SUMMARY:
The goal of this observational study is to learn about the effects of the duration of ethanol contact with the corneal surface. The main question it aims to answer is: Does this affect the behavior of corneal epithelial healing?

DETAILED DESCRIPTION:
The study was carried out on 70 patients who were candidates for laser corneal refractive surgery with alcohol-assisted PRK. The study comprised two groups. Group 1 included the right eye of the patients, and Group 2 included the left eye of the same patients. Group 1 was operated with PRK with alcohol 20% applied for 15 seconds, while group 2 underwent PRK with alcohol 20% applied for 30 seconds. Mitomycin C (MMC) 0.02% was applied for 30 seconds after the laser ablation in both groups.

Inclusions criteria:

The included patients should meet the following criteria: age between 18 and 35 years, both genders, with normal corneal topography, clear cornea, and stable refractive error for at least 12 months before the surgery. Both eyes should have low to moderate myopia with spherical error of more than -4D spherical error, cylindrical error of more than -1.5D, and an estimated stromal ablation depth of less than 70 µm.

Exclusion criteria:

The patients were excluded from the study if they had one or more of the following findings: patients with mixed astigmatism in either eye, contact lens wearers, abnormal corneal topography, thin cornea less than 500 microns, corneal opacity, dry eye disease, history of herpetic keratitis, corneal epithelial pathology (dystrophies or scarring), atopy, collagen diseases, autoimmune disease, systemic diseases that interfere with healing (e.g. diabetes mellitus), eyelid diseases, ocular pathology, previous history of refractive or corneal surgery, and pregnant or lactating females. Also, patients who failed to attend the follow-up visits were excluded.

Preoperative assessment The following preoperative measurements and examinations were performed. Uncorrected visual acuity (UCVA) and best-corrected visual acuity (BCVA) using Snellen's charts. Manifest and cycloplegic refractions were measured with the autorefractor/keratometer. Intraocular pressure measurement was done using the I Care Tonometer. Clinical examination with the slit-lamp biomicroscopy, including dilated fundus examination of the posterior segment. Then patients were examined with Pentacam HR (Oculus Optikger- ate GmbH, Wetzlar, Germany) for corneal assessment and with I design for higher order aberration measurement.

Operative details:

Preoperatively, antibiotic (Moxifloxacin hydrochloride 0.5%) and anesthetic (benoxinate hydrochloride 0.4%) eye drops were instilled on the corneal surface. Povidone-iodine 5% solution was used for sterilization, and an eyelid closed loop speculum was used to keep the eyes wide open during the procedure.

Epithelial removal was done with a sponge soaked in a 20% ethanol solution applied on the central corneal surface for 15 seconds in the right eye (group 1) and for 30 seconds in the left eye (group 2) of the same patient. Then, the corneal surface was flushed with a balanced salt solution (BSS) to remove alcohol remnants. This was followed by epithelial delamination with a dry cellulose sponge to debride an 8 mm area. A blunt spatula was used to complete this step if epithelial removal was difficult with the sponge.

Subsequently, customized PRK was performed on the dry Bowman's layer surface by VISX star S4™ excimer laser [Abbott Medical Optics Inc. (AMO), Santa Ana, CA, USA]. The targeted postoperative refraction was emmetropia for all patients.

The patients were treated with topical instillation of antibiotic drops (gatifloxacin 0.5%) four times daily for one week, topical instillation of steroid drops (prednisolone 1%) four times daily for 2 weeks, then 3 times for 2 weeks, At the second month, prednisolone was substituted by fluorometholone (0.1%) drops for 2 weeks& artificial tear drops (sodium hyaluronate 0.2%) five times daily for 3-months. An adjuvant therapy was added to the standard treatment regimen to augment the epithelial healing process: vitamin C 500 mg capsules twice per day & vitamin A 50.000 I.U. capsules once per day, both for 2 weeks.

All patients were examined daily until complete epithelial healing, then after 1 week and 3 weeks. Contact lenses were removed for all patients after 7 days.

Pain assessment:

The patients recorded their pain using a validated numerical rating scale (NRS), where the patients subjectively rated their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst imaginable pain).16

ELIGIBILITY:
Inclusion Criteria:

* The included patients should meet the following criteria: age between 18 and 35 years, both genders, with normal corneal topography, clear cornea, and stable refractive error for at least 12 months before the surgery. Both eyes should have low to moderate myopia with spherical error of more than -4D spherical error, cylindrical error of more than -1.5D, and an estimated stromal ablation depth of less than 70 µm.

Exclusion Criteria:

* The patients were excluded from the study if they had one or more of the following findings: patients with mixed astigmatism in either eye, contact lens wearers, abnormal corneal topography, thin cornea less than 500 microns, corneal opacity, dry eye disease, history of herpetic keratitis, corneal epithelial pathology (dystrophies or scarring), atopy, collagen diseases, autoimmune disease, systemic diseases that interfere with healing (e.g. diabetes mellitus), eyelid diseases, ocular pathology, previous history of refractive or corneal surgery, and pregnant or lactating females. Also, patients who failed to attend the follow-up visits were excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients seeking refarctive surgery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
epithelial healing | The patients were folllowed daily upto 2 weeks
  assessment of the time at which corneal epithelium is completely healed after PRK surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Omar, MD, Principal Investigator — Associate professor of Ophthalmology
Locations (1):
- Roaa Eye Center, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
It will be shared only on request from the principal investigator

REFERENCES:
- [Result] Goodman GL, Trokel SL, Stark WJ, Munnerlyn CR, Green WR. Corneal healing following laser refractive keratectomy. Arch Ophthalmol. 1989 Dec;107(12):1799-803. doi: 10.1001/archopht.1989.01070020881031. PMID 2597070